CLINICAL TRIAL: NCT02327351
Title: Phase II/III Study of Allogeneic Hematopoietic Stem Cell Transplantation From Unrelated and Haploidentical Donors After TCR Alfa Beta Negative Selection in Pediatric Patients With Primary Immunodeficiency Diseases
Brief Title: TCR Alpha/Beta Depletion for HSCT From Haploidentical and Unrelated Donors in the Treatment of PID
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCRabPID-2012
Record Dates: First submitted 2014-12-18; First posted 2014-12-30 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Primary Immune Deficiency Disorder; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TCR alfa beta depletion (Experimental): TCR alfa beta depleted graft, infusion. The leukapheresis product will undergo TCR alfa beta depletion following the standardized protocol.
  Interventions: Other: Biological: TCR alfa beta T cell depletion

INTERVENTIONS:
Other: Biological: TCR alfa beta T cell depletion

SUMMARY:
Treatment Study to assess of safety and efficiency of T cells receptor (TCR) alfa beta depleted graft for hematopoietic stem cell transplantation (HSCT) from haploidentical and unrelated donors in patients with primary immunodeficiency diseases

DETAILED DESCRIPTION:
Infections, graft versus host diseases (GVHD) and associated morbidity and mortality remains significant problems after unrelated and haploidentical hematopoietic stem sell transplantation (HSCT) in patients with primary immunodeficiency diseases (PID). In this study the hypothesis is that the transplantation of TCR alfa beta depleted peripheral blood stem cells (PBSC) would offers advantages over the use of positively selected CD34+ stem cells in haploidentical HSCT and non-manipulated graft in unrelated HSCT.

The purpose of this study is to evaluate the safety and efficiency of the selective infusion of TCR alfa beta T cell depleted graft in pediatric patients with PID receiving HSCT from haploidentical and unrelated donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 1 months and < 19 years
* Patients diagnosed with Primary Immunodeficiency Diseases eligible for an allogeneic transplantation and lacking a related HLA-matched donor
* Lansky/Karnofsky score > 40, WHO > 4
* Signed written informed consent

Exclusion Criteria:

* Dysfunction of liver (ALT/AST > 5 times normal value, or bilirubin > 3 times normal value), or of renal function (creatinine clearance < 30 ml / min)
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction <40%)
* Serious concurrent uncontrolled medical disorder
* Pregnant or breast feeding female patient
* Lack of parents' informed consent.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Maschan, Professor, Study Chair — Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology; Dmitry Balashov, MD, PhD, Principal Investigator — Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology
Locations (1):
- Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology, Moscow, Russia

REFERENCES:
- [Derived] Balashov D, Shcherbina A, Maschan M, Trakhtman P, Skvortsova Y, Shelikhova L, Laberko A, Livshits A, Novichkova G, Maschan A. Single-Center Experience of Unrelated and Haploidentical Stem Cell Transplantation with TCRalphabeta and CD19 Depletion in Children with Primary Immunodeficiency Syndromes. Biol Blood Marrow Transplant. 2015 Nov;21(11):1955-62. doi: 10.1016/j.bbmt.2015.07.008. Epub 2015 Jul 15. PMID 26187864

RESULTS

PARTICIPANT FLOW:
Groups:
- TCR Alfa Beta Depletion: TCR alfa beta depleted graft, infusion. The leukapheresis product will undergo TCR alfa beta depletion following the standardized protocol.
  Biological: TCR alfa beta T cell depletion
Period: Overall Study
Arm/Group | TCR Alfa Beta Depletion
Started | 98
Completed | 98
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TCR Alfa Beta Depletion
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 98
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.2 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 98

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The probability of overall survival estimated by the Kaplan-Meier method at 1 year after HSCT
Time Frame: 1 year after HSCT
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Groups:
- Matched Unrelated Donor: type of HSCT donor - HLA-matched unrelated donor
- HLA-mismatched Related Donor: type of HSCT donor - HLA-mismatched related
Arm/Group | TCR Alfa Beta Depletion | Matched Unrelated Donor | HLA-mismatched Related Donor
Number analyzed (Participants) | 98 | 75 | 23
percentage of survival probability | 86 [79 to 94] | 86 [79 to 94] | 87 [73 to 100]
Statistical Analysis 1: Comparison: Matched Unrelated Donor vs HLA-mismatched Related Donor; Test type: Superiority; p = 0.95, Gray test; survival distribution function = 86, 95% CI 2-sided [79 to 94]

2. Secondary Outcome: Transplant Related Mortality (TRM)
Description: transplant-related mortality estimated with cumulative incidence curve, considering relapse as a competitive risk
Time Frame: 24 months after transplantation
Measure: Number (95% Confidence Interval); unit: percentage of cumulative incidence
Arm/Group | TCR Alfa Beta Depletion
Number analyzed (Participants) | 98
percentage of cumulative incidence | 11 [6 to 21]

3. Secondary Outcome: Acute Graft Versus Host Diseases (аGVHD)
Description: incidence of aGVHD II-IV stage estimated with cumulative incidence curve, considering graft rejection and death as competitive risks
Time Frame: 12 months after transplantation
Measure: Number (95% Confidence Interval); unit: percentage of cumulative incidence
Arm/Group | TCR Alfa Beta Depletion
Number analyzed (Participants) | 98
percentage of cumulative incidence | 17 [1 to 28]

4. Secondary Outcome: Chronic Graft Versus Host Diseases (cGVHD)
Description: incidence of cGVHD estimated with cumulative incidence curve, considering graft rejection and death as competitive risks
Time Frame: 1 year after HSCT
Measure: Number (95% Confidence Interval); unit: percentage of cumulative incidence
Arm/Group | TCR Alfa Beta Depletion
Number analyzed (Participants) | 98
percentage of cumulative incidence | 9 [4 to 19]

5. Secondary Outcome: Cellular Immunological Reconstitution
Description: Number of participants, who reached immune recovery - CD19+ lymphocytes subsets
Time Frame: 2 years after HSCT
Population: alive at a time-point 2 years after HSCT
Measure: Count of Participants; unit: Participants
Arm/Group | TCR Alfa Beta Depletion
Number analyzed (Participants) | 70
Participants | 67

6. Secondary Outcome: Percentage of Patients With Full Donor Chimerism
Description: Percentage of patients with full (more than 90%) donor chimerism among survivals
Time Frame: last follow-up
Population: survivals at the last folow-up
Measure: Count of Participants; unit: Participants
Arm/Group | TCR Alfa Beta Depletion
Number analyzed (Participants) | 72
Participants | 48

7. Secondary Outcome: Viral Infections After Transplant
Description: number of patients with CMV reactivation (detection of any grade of CMV viremia after HSCT)
Time Frame: 12 months after transplantation
Measure: Number (95% Confidence Interval); unit: percentage of cumulative incidence
Groups:
- Matched Unrelated Donor: donor type - HLA-matched unrelated donor
- Mismatched Related Donors: donor type - HLA-mismatch relative
Arm/Group | Matched Unrelated Donor | Mismatched Related Donors
Number analyzed (Participants) | 74 | 20
percentage of cumulative incidence | 50 [38 to 65] | 60 [42 to 86]
Statistical Analysis 1: Comparison: Matched Unrelated Donor vs Mismatched Related Donors; Test type: Superiority; p = 0.35, Log Rank

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TCR Alfa Beta Depletion
All-Cause Mortality (participants affected / at risk) | 13/98
Serious Adverse Events (participants affected / at risk) | 17/98
Other Adverse Events (participants affected / at risk) | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TCR Alfa Beta Depletion (N=98)
CMV pneumonia (Respiratory, thoracic and mediastinal disorders) | 6
ADV hepatitis (Hepatobiliary disorders) | 2
Bacterial sepsis (Blood and lymphatic system disorders) | 7
TMA (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02327351/Prot_SAP_000.pdf